CLINICAL TRIAL: NCT01127724
Title: Influence of Different Doses of the Vitamin B12 on Recurrent Aphthous Stomatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties in recruiting participants
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMC105709KCTIL
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2013-04

CONDITIONS: Recurrent Aphthous Stomatitis
Keywords: Vitamin B12; Aphthous stomatitis; Cobalamin; Doses
MeSH Terms: conditions — Stomatitis, Aphthous | interventions — Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group 1- 1000 mcg (Experimental): Group I- will receive sublingual vitamin B12 treatment, 1000 mcg per day for 6 months
  Interventions: Drug: vitamin B12 treatment
- Group 2- 100 mcg (Experimental): Group II- will receive sublingual vitamin B12 treatment, 100 mcg per day for 6 months
  Interventions: Drug: vitamin B12 treatment
- group 3- 2000 mcg (Experimental): Group III- will receive sublingual vitamin B12 treatment, 2000 mcg per day for 6 months
  Interventions: Drug: vitamin B12 treatment

INTERVENTIONS:
Drug: vitamin B12 treatment — Group I- will receive sublingual vitamin B12 treatment, 1000 mcg per day for 6 months Group II- will receive sublingual vitamin B12 treatment, 100 mcg per day for 6 months Group III- will receive sublingual vitamin B12 treatment, 2000 mcg per day for 6 months
  Other Names: vitamin B12

SUMMARY:
Background: The frequency of recurrent aphthous stomatitis (RAS), the most common oral mucosa lesions seen in primary care, is up to 25% in the general population. Sublingual vitamin B12 treatment, 1000 mcg per day for 6 months was found to be effective for patients suffering from RAS, regardless of the serum vitamin B12 level. However, the optimal therapeutic dose of vitamin B12 treatment remains unclear.

Working hypothesis and aims:

Aim-To assesses the influence of different vitamin B12 treatment doses on the frequency and severity of RAS episodes.

Working hypothesis- The group receiving the higher dose of vitamin B12 treatment will have the lower frequency and severity of RAS episodes; the reaction will be faster.

Methods: randomized, double blind, intervention study.

Study population: 75 patients in three groups (total of 225 patients):

Group I- will receive sublingual vitamin B12 treatment, 1000 mcg per day for 6 months Group II- will receive sublingual vitamin B12 treatment, 100 mcg per day for 6 months Group I- will receive sublingual vitamin B12 treatment, 2000 mcg per day for 6 months Study design: Study participates will be followed through three study periods: The first period- three months prior to receiving active treatment, the second period- six month of active treatment (with randomization to study groups), and the third period- three month after finishing active treatment. Frequency and severity of RAS episodes will be recorded by the patient with "aphthous diary" that will be filled daily during all study period (12 months).

Expected results: This study will allow us to identify optimal dose of vitamin B12 treatment that will achieve faster and longer remission of RAS episodes.

Importance: This is a very common problem in the population. Study results will help to identify optimal doses of vitamin B12 needed to treat RAS.

Probable implications to Medicine: study results are supposed to give faster and better treatment for RAS episodes

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and older
* Suffer from RAS For at least one year, with aphthous frequency at least once a month.

Exclusion Criteria:

* known sensitivity to vitamin B12
* Don't speak Hebrew, Russian or English.
* Systemic Diseases, known in developing mouth aphthous (Behcet disease, Lupus Erythematosus, rheumatoid arthritis and AIDS disease)
* Patients who have received last year any form of vitamin B12 .
* Patients who receive a different treatment to RAS(not for pain)
* Pregnant or breastfeeding women
* patient suffering from Leber's optic atrophy
* Patients who suffer from Psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
frequency of recurrent aphthous stomatitis (RAS) | 12 months

SECONDARY OUTCOMES:
severity of recurrent aphthous stomatitis (RAS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yan Press, MD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Clalit Health Service (HMO), Beersheba, Israel